CLINICAL TRIAL: NCT03622515
Title: Xuanwu Hospital Capital Medical University
Brief Title: the Research of the Cerebral Protection Effects of Electroencephalogram (SedLine) During Carotid Endarterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Municipal Administration of Hospitals (Other Government)
Responsible Party: Principal Investigator, XU Na, Principal Investigator, Beijing Municipal Administration of Hospitals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZYLX201818
Record Dates: First submitted 2018-07-29; First posted 2018-08-09 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Transient Ischemic Attack; Acute Stroke; Postoperative Delirium; Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Ischemic Attack, Transient; Stroke; Emergence Delirium; Postoperative Cognitive Complications | interventions — Cerebrovascular Circulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Experimental): Sedline monitoring Adjust the depth of anesthesia by adjusting the amount of anesthesia, and adjust the cerebral perfusion pressure by adjusting blood pressure
  Interventions: Combination Product: Anesthesia level and cerebral perfusion pressure
- Group C (No Intervention): Bispectral index (BIS)/Sedline monitoring

INTERVENTIONS:
Combination Product: Anesthesia level and cerebral perfusion pressure — Anesthetic dose and blood pressure
  Arms: Group S

SUMMARY:
Fragile brain is the most common phenomenon seen in the patients undergoing CEA. The patients with fragile brain have a high incidence of postoperative brain dysfunction. This study intends to apply EEG monitoring (Sedline) to CEA to investigate whether EEG monitoring can reduce the incidence of postoperative neurological complications in CEA patients and improve their prognosis.

220 patients with CEA were randomly divided into 2 groups. Group S [Sedline monitoring + Transcranial Doppler (TCD) + regional cerebral oxygen saturation (rS02)，n=110] and group C [Bispectral index (BIS)/Sedline monitoring + TCD +rSO2,n=110], recording intraoperative and postoperative conditions, neuropsychology scale assessment, blood examination and imaging examination. The incidence of postoperative neurological complications was compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective carotid endarterectomy;
2. All those who agree to join the trial and sign the informed consent form;
3. ASAI to III.

Exclusion Criteria:

1. Those who refuse to sign the informed consent form;
2. ASA Level IV and above;
3. Unstable angina or acute myocardial infarction within 4 to 6 weeks before surgery, and heart function NYHA III to IV;
4. Those with severe liver and kidney function diseases;
5. Preoperative combined cognitive impairment; [MMSE reference demarcation value: illiterate (uneducated) group ≤ 19 points, primary school (education years ≤ 6 years) group ≤ 22 points, secondary school or above (education years) 6 years) group ≤26 points; MoCA reference demarcation value: illiterate ≤13, primary school ≤19, middle school and above ≤24. ]
6. Preoperative combined anxiety and depression; (SDS or SAS>41 points)
7. Patients with an endotracheal intubation returning to the ICU;
8. severe allergic reactions, major bleeding, etc. during surgery, causing severe fluctuations in hemodynamics;
9. The subject actively requested to withdraw from the study or to be lost to follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2018-08-10 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-04-12 (Estimated)

PRIMARY OUTCOMES:
the change from baseline of neurological complications before operation | after operation
  Transient ischemic attack, acute stroke, postoperative delirium, postoperative cognitive dysfunction, etc.

SECONDARY OUTCOMES:
the change from baseline of other complications before operation | 3 days after operation
  acute myocardial infarction, heart failure, arrhythmia, pulmonary infection, atelectasis, acute kidney injury, etc.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Xuanwu hospital Captial Medical University, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xu N, Li LX, Wang TL, Jiao LQ, Hua Y, Yao DX, Wu J, Ma YH, Tian T, Sun XL. Processed Multiparameter Electroencephalogram-Guided General Anesthesia Management Can Reduce Postoperative Delirium Following Carotid Endarterectomy: A Randomized Clinical Trial. Front Neurol. 2021 Jul 12;12:666814. doi: 10.3389/fneur.2021.666814. eCollection 2021. PMID 34322079